CLINICAL TRIAL: NCT07154992
Title: Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Efficacy and Safety of Lacticaseibacillus Rhamnosus CRL1505 in the Prevention of Upper Respiratory Tract Infections in a Healthy Paediatric Population
Brief Title: Clinical Trial to Evaluate the Efficacy of Lacticaseibacillus Rhamnosus CRL1505 in the Prevention of Upper Respiratory Tract Infections in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bioithas SL (Industry)
Collaborators: Centro Sperimentale del Latte S.r.l. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRESP.PROB-2
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Upper Respiratory Tract Infection; Prevention
Keywords: prevention; upper respiratory tract infections; probiotics; microbiota; microbiome; children
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROBIOTIC (Experimental)
  Interventions: Dietary Supplement: Probiotic - Lacticaseibacillus rhamnosus CRL1505
- PLACEBO (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic - Lacticaseibacillus rhamnosus CRL1505 — The probiotic product is provided in 2g sticks containing the strain Lacticaseibacillus rhamnosus CRL1505 at a concentration of ≥ 1.0E+8 CFU/g, with corn starch and maltodextrin as excipients.
  Arms: PROBIOTIC
Dietary Supplement: Placebo — The placebo product is provided in 2g sticks of corn starch and maltodextrin.
  Arms: PLACEBO

SUMMARY:
Randomized, double-blind, placebo-controlled, parallel-group, clinical trial to assess the efficacy of the intake of a probiotic product composed of Lacticaseibacillus rhamnosus CRL1505 strain in reducing or preventing upper respiratory tract infections (URTIs) in a healthy paediatric population.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled, parallel-group, clinical trial.

The study aims to demonstrate the efficacy of the intake of a probiotic product composed of Lacticaseibacillus rhamnosus CRL1505 strain in reducing or preventing upper respiratory tract infections in a healthy paediatric population.

The clinical trial has an intervention period of 12 weeks and a post-treatment follow-up period of 4 additional weeks (16 weeks in total).

The study aims to demonstrate the efficacy and safety of consuming the probiotic strain Lacticaseibacillus rhamnosus CRL1505 in the prevention and reduction of the severity and duration of URTI (upper respiratory tract infections) episodes in a healthy paediatric population.

A total of 268 participants aged 3 to 12 years will be recruited and randomized into two treatment groups in a 1:1 ratio (134 participants in the PROBIOTIC GROUP and 134 participants in the PLACEBO GROUP). The two intervention groups will differ based on the treatment received: probiotic or placebo, both of which will have a similar appearance.

The study will focus on a healthy paediatric population; therefore, the exclusion criteria will eliminate children with significant acute or chronic diseases and those with an immunocompromised condition. Additionally, children receiving continuous pharmacological treatment or those who have consumed dietary supplements that could influence the study results within the four weeks prior to inclusion will be excluded. However, if these children can discontinue such treatments, they may participate in the clinical trial after a washout period. Continuous regular medication that is deemed not to influence the study outcomes regarding the efficacy of the investigational product will be allowed.

Participants will be required not to modify their diet or physical activity during the course of the study.

The inclusion process will take place during winter months, to ensure that the study coincides with the months of highest URTI incidence.

Since this clinical trial will be conducted in minors, continuous evaluation will be the responsibility of the parents. They will be instructed to complete an online questionnaire daily, which will allow data collection to assess the efficacy and safety variables.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 3 to 12 years.
* Signed Informed Consent by the parents

Exclusion Criteria:

* Chronic pathological conditions, such as chronic respiratory diseases (asthma, chronic bronchitis, etc.), chronic heart diseases, chronic neurological diseases (psychomotor impairment, etc.), chronic liver diseases, chronic kidney diseases, chronic gastrointestinal diseases, hematological disorders, etc., or any other disease or condition that the investigator considers to significantly affect the health of the participating child.
* Metabolic disorders, such as diabetes mellitus, obesity, etc.
* Immunodeficiency, including HIV infection, chronic corticosteroid treatment, etc.
* Nasal polyps, nasal ulcers, or other conditions that may cause nasal obstruction.
* Regular use of medications or dietary supplements that may influence the study outcomes (immunosuppressants/immunostimulants, including echinacea supplements, analgesics, anti-inflammatory drugs, antitussives/expectorants, flu preparations, decongestants, antibiotics, antihistamines, probiotics, etc.) within the 4 weeks prior to the start of the clinical trial.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 268 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Patients who were diagnosed with at least 1, 2 or 3 URTIs | 12 and 16 weeks
  Difference in the proportion of patients who were diagnosed with at least 1, 2 or 3 URTIs during the intervention (12 weeks) and follow-up period (16 weeks) between the study groups
Number of URTIs per patient | 12 and 16 weeks
  Difference in the mean number of URTIs per patient between the study groups during the intervention period (12 weeks) and follow-up period (16 weeks)
Patients who were diagnosed of common cold and influenza | 12 and 16 weeks
  Difference in the proportion of patients who were diagnosed of common cold and influenza during the intervention (12 weeks) and follow-up period (16 weeks) between the study groups.
  *This analysis will only be performed if a considerable number of URTIs other than the common cold are recorded.

SECONDARY OUTCOMES:
Participants who presented URTI complications | 12 and 16 weeks
  Difference in the proportion of participants who experienced URTI complications (bacterial superinfections such as pneumonia, otitis media, and acute sinusitis) during the intervention period (12 weeks) and the total follow-up period (16 weeks) between the study groups.
Number of days with a URTI episode per participant | 12 and 16 weeks
  Difference in the average number of days with a URTI episode per participant (days with URTI/participants) during the intervention period (12 weeks) and the total follow-up period (16 weeks) between the study groups.
Number of days until the first URTI | 12 weeks
  Difference in the average number of days until the onset of the first URTI episode during the intervention period (12 weeks) between the study groups.
Duration of each URTI episode | 12 and 16 weeks
  Difference in the average duration of each URTI episode (mean ratio of days with URTI/URTI episodes for each participant) during the intervention period (12 weeks) and the total follow-up period (16 weeks) between the study groups.
URTI-free time rate | 12 and 16 weeks
  Difference in the URTI-free time rate (proportion of accumulated days in which participants do not experience URTI relative to the total number of days) during the intervention period (12 weeks) and the total follow-up period (16 weeks) between the study groups.
Score of each symptom evaluated on the Jackson scale | 12 and 16 weeks
  Difference in the average score of each symptom evaluated on the Jackson scale per day of common cold episode during the intervention period (12 weeks) and the total follow-up period (16 weeks) between the study groups.
  The Jackson scale (also known as Jackson criteria or Jackson score) is a tool used to assess and quantify the symptoms of upper respiratory tract infections (URTI), such as the common cold
  It evaluates 8 main symptoms:
  Sneezing, Nasal discharge (runny nose), Nasal congestion, Sore throat, Cough, Headache, Malaise, Chilliness/feverishness
  Each symptom is scored on a 0-3 scale:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe
  Criteria for defining a "cold episode" (URTI case) according to Jackson:
  At least 2 consecutive days with ≥2 of the following symptoms: runny nose, sore throat, sneezing. Or 1 of these symptoms plus at least one systemic symptom (headache, malaise, chilliness/feverishness).
Number of days with fever per participant | 12 and 16 weeks
  Difference in the average number of days with fever per participant during the intervention period (12 weeks) and the total follow-up period (16 weeks) between the study groups.
Participants who received antibiotic treatment | 12 and 16 weeks
  Difference in the proportion of participants who received antibiotic treatment during the intervention period (12 weeks) and the total follow-up period (16 weeks) between the study groups.
Number of days with antibiotic treatment per participant | 12 and 16 weeks
  Difference in the average number of days with antibiotic treatment per participant during the intervention period (12 weeks) and the total follow-up period (16 weeks) between the study groups.
Proportion of URTI episodes in which participants received symptomatic medication | 12 and 16 weeks
  Difference in the proportion of URTI episodes in which participants received symptomatic medication (to relieve URTI symptoms) during the intervention period (12 weeks) and the total follow-up period (16 weeks) between the study groups.
Proportion of URTI days in which participants received symptomatic medication | 12 and 16 weeks
  Difference in the proportion of URTI days in which participants received symptomatic medication (to relieve URTI symptoms) during the intervention period (12 weeks) and the total follow-up period (16 weeks) between the study groups.
Participants who experienced gastrointestinal infections | 12 and 16 weeks
  Difference in the proportion of participants who experienced gastrointestinal infections during the intervention period (12 weeks) and the total follow-up period (16 weeks) between the study groups.
School absence rate | 12 and 16 weeks
  Difference in the school absence rate (proportion of accumulated school absence days due to URTI relative to the total number of days) during the intervention period (12 weeks) and the total follow-up period (16 weeks) between the study groups.

OTHER OUTCOMES:
Incidence and severity of all Adverse Events | 12 and 16 weeks
  * Incidence and severity of all Adverse Events.
  * Incidence of Severe Adverse Events.
  * Incidence and severity of Adverse Events related to the study product.
  * Incidence and severity of Adverse Events leading to study withdrawal.
  * Rate of withdrawal due to intolerance to study product.

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Taverniti, Study Director — Microbes & Health R&D Leader, Centro Sperimentale del Latte S.r.l.
Locations (1):
- MiBioPath Research Group (UCAM), Murcia, Spain